CLINICAL TRIAL: NCT05843513
Title: Tooth Wear Monitoring Using Intraoral Scanner. Identification of Etiological Factors and Patient Satisfaction.
Brief Title: Tooth Wear Monitoring Using Intraoral Scanner
Status: Completed | Type: Observational
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Díaz-Flores García, Principal Investigator, Universidad Europea de Madrid
Other Study IDs: Desgaste-UE
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Dental Wear
Keywords: Dental wear; Intraoral scanner; Etiological factors; Monitoring
MeSH Terms: conditions — Tooth Wear | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Monitoring: From every participant the following information was recorded for further analysis:
  * State Trait Anxiety Inventory (STAI) questionnaire.
  * A questionnaire is carried out to assess:
    1. Endogenous abrasion: presence or absence of wear facets; carrier of occlusal splint; presence of harmful oral habits; day and/or night grinding.
    2. Exogenous abrasion: whether they bite hard or soft things.
    3. Exogenous erosion: - Environmental factors: frequent swimming. - Ingestion of acidic drinks or substances: fizzy drinks, juices, alcohol, dressings, etc.
    4. Endogenous erosion: reflux, vomiting, heartburn, nighttime drooling, etc.
  * An examination of the temporomandibular joint (TMJ) is carried out; palpation of the muscles most frequently related to bruxism and/or alterations of the TMJ.
  * 2 Intra oral scans (IOS): Baseline and follow up (1 year after baseline) to perform a quantification of tissue loss (over 100 microns) using Geomagic software.
  Interventions: Other: Monitoring (observational study)

INTERVENTIONS:
Other: Monitoring (observational study) — The relationship between dental wear and the behaviour of the participants will be analysed.

SUMMARY:
The overall objective was to evaluate the monitoring of tooth wear using the intraoral scanner. Forty-six participants were selected according to the established inclusion and exclusion criteria. Monitoring of tooth wear, evaluation of possible aetiological factors, as well as patient satisfaction with the use of the intraoral scanner were carried out.

DETAILED DESCRIPTION:
The overall objective was to evaluate the monitoring of tooth wear using the intraoral scanner. The specific objectives were (1) to determine whether the intraoral scanner is capable of detecting tooth wear superior to traditional visual indices, (2) to identify whether any aetiological factors may be associated with tooth tissue loss, (3) to establish a degree of patient satisfaction with the intraoral scanner as a diagnostic tool. Forty-six participants were selected according to the established inclusion and exclusion criteria. The protocol was accepted by the Regional Ethics Committee of the Community of Madrid. Digitisation of the dental arches was recorded at 3 types of evaluation: 0, 6 months and 12 months. The recording of possible etiologic factors was carried out at the three established evaluation times. The evaluation of satisfaction was recorded at the third evaluation time.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age
* patients who were to stay at the university for more than one and a half years
* patients who agreed to sign the informed consent form.

Exclusion Criteria:

* pregnant women
* patients who planned to modify the oral situation with orthodontic, surgical and/or rehabilitative treatments
* patients who had some kind of personal or academic relationship with the investigators of this study.

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Adults between 18 to 40.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Tooth wear monitoring | 1 year
  Quantification of tissue loss (more than 100 microns) using intraoral scanner related with possible etiological factors

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garcia VD, Freire Y, Fernandez SD, Murillo BT, Sanchez MG. Application of the Intraoral Scanner in the Diagnosis of Dental Wear: An In Vivo Study of Tooth Wear Analysis. Int J Environ Res Public Health. 2022 Apr 8;19(8):4481. doi: 10.3390/ijerph19084481. PMID 35457351
- [Result] Travassos da Rosa Moreira Bastos R, Teixeira da Silva P, Normando D. Reliability of qualitative occlusal tooth wear evaluation using an intraoral scanner: A pilot study. PLoS One. 2021 Mar 25;16(3):e0249119. doi: 10.1371/journal.pone.0249119. eCollection 2021. PMID 33765042